CLINICAL TRIAL: NCT02171247
Title: Comparison of the Use of High Iodine Concentration Contrast Material (Isovue 370) vs. Standard Protocol in Coronary Computed Tomographic Angiography (CTA)
Brief Title: Comparison of Isovue 370 vs. Standard Protocol in Coronary Computed Tomographic Angiography (CTA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00004492
Record Dates: First submitted 2014-06-12; First posted 2014-06-24 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Coronary Computed Tomographic Angiography
Keywords: coronary computed tomographic angiography; contrast
MeSH Terms: interventions — Iopamidol

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Isovue 370 (Active Comparator): Isovue 370 is a contrast agent with increased iodine concentration.
  Interventions: Drug: Isovue 370
- Visipaque 320 (Active Comparator): Standard protocol is Visipaque 320.
  Interventions: Drug: Visipaque 320

INTERVENTIONS:
Drug: Isovue 370 — Isovue 370 is a contrast agent with increased iodine concentration.
  Arms: Isovue 370
Drug: Visipaque 320 — Visipaque 320 is standard protocol.
  Arms: Visipaque 320

SUMMARY:
Computed Tomography Angiogram (CTA) scans are performed routinely to look at the vessels in the body as an alternative to directly injecting contrast into the vessels and taking pictures. Different types of intravenous (into the vein, IV) contrast are available to fill the vessels and make them easier to see. The purpose of the study is to determine the best type of contrast for this scan.

ELIGIBILITY:
Inclusion Criteria:

* adult patients who are referred for coronary CTA for suspected or known coronary artery disease

Exclusion Criteria:

* creatinine greater than 2.0
* allergy to contrast media
* patients under the age of 18
* women who are pregnant or breast feeding
* patients with cardiac arrhythmia will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T Boll, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 subjects signed consent. 2 subjects were not assigned to a arm and were withdrawn from study due to impaired renal function. 33 subjects completed the study.
Period: Overall Study
Arm/Group | Visipaque 320 | Isovue 370
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Visipaque 320 | Isovue 370 | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Customized [Number; unit: participants]
  18 years and older | 16 | 17 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Contrast to Noise Ratio
Description: Contrast-to-noise ratios (CNRs) were calculated as follows: CNR = (vascular attenuation - myocardium attenuation) / SD of mean noise attenuation.
Time Frame: during scan, approximately 3 hours
Measure: Mean (Standard Deviation); unit: CNR
Arm/Group | Visipaque 320 | Isovue 370
Number analyzed (Participants) | 16 | 17
CNR | 18.6 (5.2) | 20.5 (4.5)

2. Primary Outcome: Image Quality
Description: Depiction of Branch Vessels - coronary branch depiction was performed as consensus decisions of two blinded radiologists. Criteria used was abscence or presence of vessels.
Time Frame: during scan, approximately 3 hours
Measure: Number; unit: % of coronary branches visualized
Arm/Group | Visipaque 320 | Isovue 370
Number analyzed (Participants) | 16 | 17
% of coronary branches visualized
  Conus | 43.8 | 94.1
  Sinoatrial Nodal | 37.5 | 82.4
  Diagonal1 | 87.5 | 35.3
  Diagonal1 and Diagonal2 | 12.5 | 64.7
  Obutse Marginal1 | 68.8 | 29.4
  Obutse Marginal1 and Obutse Marginal2 | 6.3 | 70.6
  Acute marginal1 | 62.5 | 47.1
  Acute marginal1 and Acute marginal2 | 18.8 | 52.9
  Septal perforator | 43.8 | 88.2
  Posterolateral | 6.3 | 64.7

3. Primary Outcome: Motion Artifact
Description: The outcome will be measured by individual scores. The scores from multiple readers will be averaged.
Time Frame: during scan, approximately 3 hours
Population: Data was not collected and therefore not analysed
Arm/Group | Visipaque 320 | Isovue 370
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Attenuation of the Ascending Aorta and Coronary Arteries
Description: The investigator will measure the length of visualized coronary artery for the left anterior descending, left circumflex and right coronary arteries as a way of quantifying visualization of distal coronary segments.
Time Frame: during scan, approximately 3 hours
Measure: Mean (Standard Deviation); unit: CNR
Arm/Group | Visipaque 320 | Isovue 370
Number analyzed (Participants) | 16 | 17
CNR
  ascending aorta | 19.5 (4.8) | 21.6 (4.2)
  coronary arteries | 18.4 (5.3) | 20.3 (4.6)

ADVERSE EVENTS:
Arm/Group | Visipaque 320 | Isovue 370
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes